CLINICAL TRIAL: NCT05702151
Title: Erector Spinae Plane Block in Robotic Cardiac Surgery
Brief Title: ESP Block in Robotic Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESProbot001
Record Dates: First submitted 2022-12-19; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-11

CONDITIONS: Heart Valve Diseases; Postoperative Pain, Acute; Analgesia
Keywords: Robotic Cardiac Surgery; ESP Block; Postoperative Pain; Heart Valve disease
MeSH Terms: conditions — Heart Valve Diseases; Pain, Postoperative; Agnosia | interventions — Morphine; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Open Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine infusion (Active Comparator): IV morphine 50mcg/kg/h infusion with Patient Controlled Analgesia extra bolus on demand of 1mg (lockout interval 20 minutes), and paracetamol 1g every 8 hours.
  Interventions: Drug: Morphine injection
- ESP Block analgesia (Experimental): After induction of anesthesia in the operating room, the patient is positioned in lateral decubitus. Under strict aseptic conditions, and guided by ultrasound, an Erector Spinae Plane block is performed injecting ropivacaine 0.2% 20ml, and a catheter is placed.
  An infusion of ropivacaine 0.16% at 10ml/h is started in the operating room. Patient Controlled Analgesia pump will be connected with 1mg IV morphine bolus on demand, and paracetamol 1g every 8 hours, is also delivered.
  Interventions: Procedure: ESP Block; Drug: Morphine injection

INTERVENTIONS:
Procedure: ESP Block — After induction of anesthesia in the operating room, the patient is positioned in lateral decubitus. Under strict aseptic conditions, and guided by ultrasound, an Erector Spinae Plane block is performed injecting ropivacaine 0.2% 20ml, and a catheter is placed. Ropivacaine 0.2% infusion at a 10ml/h rate is started during the surgery.
  Other Names: Erector spinae Plane Block
  Arms: ESP Block analgesia
Drug: Morphine injection — Intravenous morphine infusion 50mcg/kg/h with Patient Controlled Analgesia extra bolus on demand (1mg bolus with 20 minutes lockout time), and paracetamol 1g every 8 hours.
  Other Names: Intravenous opioid infusion analgesia and paracetamol

SUMMARY:
Patients undergoing cardiac robotic surgery will receive different pain management after being randomized in 2 groups. Control group will receive standard of care pain management with acetaminophen and morphine in PCA pump, and the intervention group will receive an erector spinae plane block with a continous infusion of local anesthetic.

At 3 months the patients will be contacted to assess for pain and ask them for they life quality.

DETAILED DESCRIPTION:
Patients undergoing cardiac robotic surgery will receive different pain management after being randomized in 2 groups. Before the surgery and after checking eligibility criteria and exclusion criteria the patients will be asked to enroll to the study. If the agree to participate, they will sign de informed consent and fill the EQL 5D-5L questionnaire.

The day of the surgery, the perioperative process will be performed as usual unless the interventions detailed in this description.

Patients will be transferred to the surgical area, enter to the operating room, monitored and general anesthesia will be performed.

Standard postoperative analgesia group will receive a at the end of the surgery a bolus of IV morphine 0,05mg/kg, followed with infusion of IV morphine 0,25mg/h in Patient Controlled Analgesia protocol (extra bolus on demand of 1mg with lockout interval 20 minutes), and paracetamol 1g every 8 hours.

The experimental group will receive the standard analgesia and an ESP Block. In this group, after the induction of general anesthesia in the operating room, the patient is positioned in lateral decubitus. Under strict aseptic conditions, and guided by ultrasound, an ipsilateral Erector Spinae Plane block is performed injecting ropivacaine 0.2% 20ml, and a catheter is placed in this plane.

An infusion of ropivacaine 0.16% at 10ml/h is started in the operating room.

Both groups of patients will emerge from anesthesia in the operative room or at the intensive care unit in the first 6 postoperative hours if possible. After the surgery they will be transfered to the intensive care unit where vital signs will be monitored continuously.

The pain intensity and the total required opioid dose will be registered at 12, 24 and 48 postoperative hours. After acute phase of postoperative pain and typically until chest drainages are retired, the ESP catheter and the IV morphine will be withdrawn. After discharge by usual criteria, 3 months after the surgery patients will be contacted by telephone. Quality of life, pain and if present, its characteristics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Robotic Cardiac Surgery
* Accepts to participate

Exclusion Criteria:

* Use of other regional anesthesia technics
* Presence of chronic Pain
* Psychiatric pathology, drug abuse
* Allergy or intolerance to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Accumulated opioid dose 12h | 12 postoperative hours
  Morphine PCA pump will measure the accumulated dose of morphine, this is an objective measure of how many times the patients have had uncontrolled pain. Expressed in mg. If the patient has received other opioid besides of morphine it will be transformed using equivalent morphine dose and added to the total dose.
Accumulated opioid dose 24h | 24 ostoperative hours
  Morphine PCA pump will measure the accumulated dose of morphine, this is an objective measure of how many times the patients have had uncontrolled pain. Expressed in mg. If the patient has received other opioid besides of morphine it will be transformed using equivalent morphine dose and added to the total dose.
Accumulated opioid dose 48h | 48 postoperative hours
  Morphine PCA pump will measure the accumulated dose of morphine, this is an objective measure of how many times the patients have had uncontrolled pain. Expressed in mg. If the patient has received other opioid besides of morphine it will be transformed using equivalent morphine dose and added to the total dose.
Visual Analogic Scale 12h | 12 postoperative hours
  Pain will be measured with Visual analogic scale and recorded. It has numeric discrete ranging from 0 to 10.
Visual Analogic Scale 24h | 24 postoperative hours
  Pain will be measured with Visual analogic scale and recorded. It has numeric discrete ranging from 0 to 10.
Visual Analogic Scale 48h | 48 postoperative hours
  Pain will be measured with Visual analogic scale and recorded. It has numeric discrete ranging from 0 to 10.

SECONDARY OUTCOMES:
EQ 5-Dimensions 5-Levels | Preoperative and 3 months after surgery
  Quality of Life measure with EQ 5D 5L scale, created by the Euro QL group and used to measure life quality, its a scale describing 5 dimensions of life (Mobility, Self care, General activity, pain and discomfort, anxiety and depression) in 5 levels of comfort/discomfort (Score of 1 in each dimensions describes the most comfort). It can be expressed separately or by combining them into an index generated with a standard calculator provided by the EQL group.
Brief Pain Scale | 3 months after surgery
  Pain presence and its characteristics 3 months after surgery described by the brief pain scale. This standard scale describes the pain intensity from 1 to 10 (being 10 the most intense pain) and and DN4 scale will be performed.
Neuropathic pain assessment | 3 postoperative months
  When pain is present, assessment for neuropathic pain characteristics will be assessed using the Douleur neuropathique 4 (DN4) scale, spanish version. This scale assess 10 characteristics of pain, with a maximum score of 10, minimum of 0. Interpreted as positive (neuropathic pain likely) with a score of 7 or more.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD, unless requested

REFERENCES:
- [Background] Rovira Canudas I. [Postoperatory analgesia for minimally invasive cardiac surgery: which is the ideal technique?]. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):467-9. doi: 10.1016/j.redar.2012.07.010. Epub 2012 Sep 12. No abstract available. Spanish. PMID 22980395
- [Background] Freise H, Van Aken HK. Risks and benefits of thoracic epidural anaesthesia. Br J Anaesth. 2011 Dec;107(6):859-68. doi: 10.1093/bja/aer339. Epub 2011 Nov 4. PMID 22058144
- [Background] D'Ercole F, Arora H, Kumar PA. Paravertebral Block for Thoracic Surgery. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):915-927. doi: 10.1053/j.jvca.2017.10.003. Epub 2017 Oct 4. PMID 29169795
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068